CLINICAL TRIAL: NCT03469791
Title: Less Invasive Decompression Alone as Good as Decompression Plus Instrumented Fusion for Lumbar Spinal Degenerative Spondylolisthesis at Long Term? A Pragmatic Comparative Non-inferiority Observational Study From the Norwegian Registry for Spine Surgery
Brief Title: Degenerative Spondylolisthesis; Micro-decompression vs Decompression + Instrumented Fusion; Long Term Follow up
Acronym: DS-registry
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/344
Record Dates: First submitted 2018-03-05; First posted 2018-03-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Degenerative Lumbar Spondylolisthesis
Keywords: Degenerative Spondylolisthesis; Treatment; Decompression alone; Instrumented fusion; Oswestry Disability Index

STUDY DESIGN:
Intervention Model Description: Non-inferiority cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Micro-decompression alone (Active Comparator): In Surgical treatment of Degenerative Spondylolisthesis patients are operated on with a midline-precerving decompression without fusion
  Interventions: Procedure: Surgical treatment of Degenerative Spondylolisthesis
- Decompression and instrumented fusion (Active Comparator): In Surgical treatment of Degenerative Spondylolisthesis patients are operated on with a decompression followed by an instrumental fusion with or without an additional Cage
  Interventions: Procedure: Surgical treatment of Degenerative Spondylolisthesis

INTERVENTIONS:
Procedure: Surgical treatment of Degenerative Spondylolisthesis

SUMMARY:
In many countries a majority of patients with degenerative spondylolisthesis are operated on with decompression plus instrumented fusion, but the scientific evidence for adding fusion is controversial. To evaluate whether micro-decompression alone is as good as (non-inferior to) decompression plus instrumented fusion, a study with data from the Norwegian Registry for Spine Surgery was conducted, now the long-term follow up.

DETAILED DESCRIPTION:
It is moderate evidence for that surgical treatment is superior non-surgical treatment for Degenerative Spondylolisthesis (DS). Question regarding the effectiveness of different surgical treatment alternatives is a controversy. The main goal for an operation is to decompress the stenotic neural elements. Based on two influential studies in the early1990's, an additional fusion procedure became more and more common and during the next decades the rate of fusion procedures as well as the complexity of the fusion procedures increased dramatically. In 2011 about 90 % of the surgeries performed in the United States included an instrumented fusion procedure. This practice has been supported by several guidelines and reviews. However, the evidence for this practice has been questioned and as a consequence of the conflicting results from two randomised controlled trial, the role of fusion again has become controversial.

According to the annual reports from Norwegian Spine Registry (NORspine), the majority of the decompression alone surgeries for DS is performed with preserving of the midline structures. These procedures are considered to be biomechanical less extensive and may result in less instability and less progression of the slip compared to a standard laminectomy.

In the now published Norwegian study (NORSTEN-DS; Clinicaltrial.gov Identifier: NCT02051374) DS the participants were randomised into micro-decompression alone and decompression plus instrumented fusion. In the observational non-inferiority cohort study the investigators evaluated the effectiveness of micro-decompression alone and decompression plus instrumented fusion among patients registered in the NORspine registry. The hypothesis was that the clinical result for the micro- decompression group is as good as the results for the instrumented fusion group, at short time (12 months after operation) and at long time (7 to 15 years after operation) for DS .

Statistics For the complete cohort of patients fulfilling the inclusion and exclusion criteria, the baseline demographics and outcome measures will be presented.

To as best as possible adjust for covariate that can bias the allocation to treatment, Propensity score matching (PSM) will be used to make the distribution of observed baseline patient characteristics in the micro-decompression group and the fusion group as similar as possible. The following parameters will be included in the calaculation of the propensity score: Age; Gender; American Society of Anesthesiologists (ASA) grade; Body Mass Index (BMI); Smoking, Oswestry Disability Index(ODI), Numeric Rating Scale for leg pain and for back pain, Euroqol 5-D (EQ5D), foraminal stenosis, degenerative disc disease, predominating back pain, number of levels operated on and neurological palsy. The PSM scores will be derived from a logistic regression model and reflect a patient's theoretical baseline probability for being instrumentally fused. Using the technique of '1:1 matching without replacement', pairs of fused and non-fused patients with a difference in propensity scores less than 0.2 in logit of the standard deviation will be formed.

In order to include data from all three time points and hence make use of all available data, Latent Growth Curve (LGC) models with Full Information Maximum Likelihood will be used for estimating the change scores and the follow-up scores for ODI ,NRS leg pain and NRS back pain. Thus, information from patients will not be excluded if data are missing at one of the follow-ups. Statistical Package for the Social Sciences (SPSS) version 24 will be used for descriptive statistics, tests for distribution of data, cross-tabulations with χ2 test, Student t-tests and Mann-Whitney U tests of group differences and linear and logistic regression modelling Mplus verion 7.3 will be used for analysing LGC models.

To control for biased estimate due to data missingness, a sensitivity analysis will be performed. With use of baseline and follow-up data as predictors for multiple imputation (MI), 10 data sets will be generated with complete follow-up scores for ODI, NRS leg pain and NRS back pain.

The sample size calculation for comparing the effectiveness of the treatments is based on the same assumption as the randomized multicentre trial on the same patient group (ClinicalTrials.gov Identifier: NCT02051374). In a non-inferiority design, with one sided testing, the investigators want to detect whether the responder rate for the micro-decompression group is less than 15 percentages lower than for the fusion group. This has to be tested by forming a 95% confidence interval (CI) for the difference of proportions (i.e. percentage of responders in the fusion group minus percentage of responders in the micro-decompression group) and has to be rejected if the upper limit of the CI is less than 15. If rejected, the conclusion will be that decompression alone is non-inferior, i.e. as good as, decompression with fusion. A 15% difference in responder rate corresponds to a number needed to treat of 7 patients (NNT = 100/15 = 6.67 [12]. Choosing a type 1 error = 0.05 and power = 0.90 gives a sample size of 160. Considering these assumptions, and adding 25% for possible dropouts, a total of 213 patients are required in each group.

To investigate the long term results, we will perform a similar study with data at long term follow-up (5 to 15 years postoperatively) including the same patients as in the primary study (one year follow-up). The patients will receive a similar questionnaire as used in the primary study. The design, primary outcome, secondary outcomes, hypothesis, hypothesis testing, non-inferiority margin and statistical methods will follow the same rules as for the primary study. When analyzing the clinical outcomes (patient reported outcome measurements) the statistician will be blinded for treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* operated between September 2007 and December 2015 labeled in the registry with both 'Spinal stenosis' and 'Degenerative spondylolisthesis'
* operated on with decompression with or without an additional fusion

Exclusion Criteria:

* operated with an anterior approach
* had a former operation at index Level
* was labeled with a degenerative scoliose
* was operated in more than 2 Levels
* was operated with non-instrumented fusion
* operated with a standard laminectomy with removing of the posterior midline structures or operated without magnifying devices was excluded from the micro-decompression group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2007-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Responder rate assessed by ODI | From date of operation to 12 month follow-up. From date of operation to long-term(7-15 yrs) follow-up
  The proportion of participants with an improvement on the Oswestry Disability Index score score more than 30% from preoperative to 12 month and long term follow-up.ODI is a self-reported instrument comprising 10 sections where the patient is supposed to mark the most appropriate item.The sum score range from 0 to 100 were 100 represent the greatest impairment.

SECONDARY OUTCOMES:
ODI: Mean change and mean follow-up score | From date of operation to 12 month follow-up and to long term follow-up (7 -15 yrs)
  Mean change from date of operation to 3 month follow-up, from 3 to 12 month follow-up, from 12 month to long term, the mean follow-up score at 12 month and at long term follow up.
NRS leg pain | From date of operation to 12 month follow-up and long term follow up (7-15 yrs)
  Mean change from date of operation to 3 month follow-up, from 3 to 12 month follow-up and the mean follow-up score at 12 month and long term (7-15yrs) for the Numeric Rating Scale [(NRS; which ranges from 0 to 10 (worst pain imaginable)] for leg pain.
NRS back pain | From date of operation to 12 month follow-up and long term follow up (7-15 yrs)
  Mean change from date of operation to 3 month follow-up, from 3 to 12 month follow-up and the mean follow-up score at 12 month and at long term (7-15 yrs)for NRS back pain
GPE scores | At 12 month follow-up and at long term follow up (7-15yrs)
  Global Perceived Effect scale (GPE; a global assessment of patient-rated satisfaction with treatment outcome, with the answers 'completely recovered'=6, 'much improved'=5, 'slightly improved'=4, 'unchanged'=3, 'slightly worse'=2, 'much worse'=1 and 'worse than ever'=0. The GPE-responses will be trichotomised into 'substantially improved' ('completely recovered' and 'much improved'), 'slight or no change' ('slightly improved', 'unchanged' and 'slightly worse') and 'substantially deteriorated' ('much worse' and 'worse than ever')
Hospital stay | Up to 12 months
  The length of hospital stay
Operation time | Perioperative
  The duration of surgery
Complications | From date of operation to 3 month follow-up
  The rate of perioperative complications and adverse events registered on the surgeon form and the rate of patient-reported complications and adverse events the first 3 months postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Ivar Magne Austevoll, PhD, Principal Investigator — Haukeland University Hosptal; Eric Loratang Kgomotso, MD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Kysthospitalet i Hagevik, Orthopeadic Clinic, Haukeland University Hospital, Bergen, Hagevik, Norway